CLINICAL TRIAL: NCT06812442
Title: Effectiveness of a 3-month Individual Reminiscence Therapy Program on Global Cognition, Mood, and Quality of Life in Older Adults With Mild to Moderate Alzheimer's Disease: A Multicenter Randomized Controlled Trial
Brief Title: Effectiveness of a 3-month Individual Reminiscence Therapy Program in Older Adults With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rsocialform - Geriatria, Lda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01022025
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Dementia; Alzheimer Disease; Cognitive Impairment
Keywords: older adults; reminiscence therapy; quality of life; mood; depression; anxiety; Alzheimer´s disease; non-pharmacological therapies; randomized controlled trial
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who meet the inclusion criteria will be randomly assigned to the intervention group receiving Reminiscence Therapy (RT) or to a control group receiving only Treatment as Usual (TAU). Participants in the intervention group will participate in two RT sessions per week for 13 weeks besides their TAU. The sessions will be based on the Book of the Past and the Present and they will follow the same protocol in every participant site.
  Interventions: Other: Reminiscence therapy
- Control Group (No Intervention): Participants assigned to the control group will maintain TAU in the site, participating in the activities previously assigned to their individual care plan.

INTERVENTIONS:
Other: Reminiscence therapy — Intervention group will receive two RT sessions per week for 13 weeks. RT sessions will last approximately 50 minutes and will be developed according to the following structure: · Welcome to the patient and reality orientation therapy (7 minutes)· Conducting the main activity of reminiscence (40 minutes) · Closure, thank you for the participation and farewell until the next session (3 minutes). RT sessions will have an individual format and will be conducted by a therapist previously trained in the protocol and the principles of RT. The Reminiscence activities of each session will be carried out following the protocol proposed in the Book of the Past and the Present.
  Arms: Intervention Group

SUMMARY:
This research aims to evaluate the effectiveness of individual Reminiscence Therapy (RT) program, using a simple reminiscence format, to improve the overall cognitive function, mood, and quality of life (QoL) of older adults with mild to moderate Alzheimer's disease attending social care and support services. A multicentre randomised controlled trial (RCT) is proposed in Portugal with repeated measures (pre-intervention, and post-intervention). Intervention group will hold 26 individual RT sessions, twice a week for 13 weeks. Control group participants will maintain their treatment as usual. Make a subsample analysis of the main clinical diagnoses, and compare the results of sample and subsample with a previous study that had the same intervention protocol.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a genetic and sporadic neurodegenerative disease that is associated with a decline in cognitive function, memory, speech, and ultimately sensory and motor problems. The onset of these changes may be gradual or sudden. In people with mild Alzheimer's, symptoms such as learning and memory problems, poor judgment, mood swings, depression, and restlessness occur.

The absence of an effective pharmacological treatment that halts or delays the development of the disease has aroused interest in non-pharmacological therapies (NPT) as a complement to pharmacological treatment that can improve the quality of life of older adults with AD. One of the most researched NPT and with the greatest tradition in this field is Reminiscence Therapy (RT).

RT implies the discussion of past activities, events and experiences, usually with the help of triggers (e.g., photographs, home objects and other familiar items from the past, music, any object or stimulus) that serve to stimulate memories. In its application to dementias, RT is based on the fact that the memory deficit of people with dementia implies that they are able to remember events from their past life, especially from childhood to early adulthood, but not newer facts. It focuses on preserved capacities and memories, promotes communication and enables the person to connect with his past and recover his sense of personal identity. In this way, the RT can be understood as an intervention on the edge of those of cognitive orientation and those centred on emotion, with potential interactive effects on autobiographical memory and psychological well-being.

In simplified form, there are at least two approaches to RT. The first approach as a "life review" where participants are guided through significant experiences of their biography trying to give meaning to their lives. This type of RT is more structured and is usually conducted in an individual format. It may involve the production of "life books". This approach is considered to have an integrative function aimed at achieving a sense of validation, coherence and reconciliation with one's past. Another approach that call general or simple reminiscence, implies the stimulation of autobiographical memory during conversations on specific themes of the past (e.g, holidays, food and drink, work) using stimulus to trigger memories. It has been described as an unstructured autobiographical memory narration. This reminiscence format can be conducted both individually and in groups and promotes communication between participants who share their memories and stories.

In either format that RT is applied on, the introduction of triggering stimulus (e.g., photographs, music, old objects) to help memory is considered fundamental. These triggers can be generic, reflecting common experiences in the lives of people relevant to their age group (e.g., a school manual can serve as a reminder of the experience during their school stage), or specific, with stimulus related to the person's own experiences (e.g., photographs of an important vital event such as their wedding day or a journey during their youth).

As for the effectiveness of RT, according to a review by Woods et al. in Cochrane, there is some evidence on its positive effects on cognition, QoL, communication and possibly on the mood of people with dementia, even if the benefits are small. Despite the distinction between the two different approaches to RT (general reminiscence vs. life history), the therapy modality does not seem to be as important to achieve positive effects as the individual or group format of the sessions and the context in which the intervention is administered (people living in the community or institutionalised).

In particular, according to the results of the review study, the RT seems to be able to generate a small benefit on cognitive function immediately after the intervention, although it usually does not continue after a longer follow-up period. Regarding the administration format, the individual RT seems slightly superior in its effects on cognition both immediately and after a follow-up period. In any case, its effects seem comparable to those of other cognitive stimulation modalities.

As for the effect of RT on quality of life (QoL), an individual RT study based on life review, showed an improvement in Qol-AD. The effects with a group modality do not seem consistent, showing little or no effect on QoL, although the key factor may be the context of application (community vs. institution), with better group RT results in institutionalised patients.

In a multicentre study conducted in Portugal with older adults with neurocognitive disorders, in individual format, there was a significant effect on the overall cognition, memory and QoL of the participants. Group RT was associated with a likely effect on communication both after the intervention and in the follow-up. This effect was not replicated in the individual RT, with uncertain results.

Finally, despite the evidence on the effect of RT on the mood of older adults without dementia, in the case of people with dementia only a small effect on mood was found for those participating in individual RT. In the portuguese multicentre studies there were no significant differences in depressive symptomatology.

Based on the above, this research proposal aims to evaluate the effectiveness of individual RT program within a general reminiscence format, to improve overall cognitive function, emotional state (depression and anxiety), and QoL of older adults with AD attending social care and support services in the Portugal.

It is proposed to evaluate the efficacy of the intervention in the endpoint assessment. Furthermore, an analysis of results based on the diagnosis of the participants is proposed for those diagnoses with sufficient representation in the sample (more than 15 cases in each group). Additionally, it is proposed to analyze the factors that predict the response to the intervention (responder analysis). Finally, the results of this study will be compared and can be analyzed together with those of a previous studies that used the same individual RT program and the same experimental design.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older.
* Receiving care and support services for at least three months.
* Diagnosis of probable Alzheimer's disease according to Diagnostic and Statistical Manual of Mental Disorders (DSM), fifth edition text revision criteria.
* Intact communication skills.
* Native Portuguese speaking.
* Signed informed consent by the participant.
* Mini Mental State Examination (MMSE) score between 10 and 24 points

Exclusion Criteria:

* Severe sensory and physical limitations.
* Acute or serious illness precluding participation in the RT sessions.
* Evidence of aggressive and disruptive behaviour, as observed by staff at the facility.
* Starting neuroleptics or antipsychotics within two months of recruitment.
* No literacy (educational level).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning evaluated through Mini-Mental State Examination (MMSE) | baseline
  MMSE is a widely used screening tool that evaluates cognitive domains such as orientation, attention, memory, language, and visual-spatial skills. Scores range from 0 to 30, with higher scores indicating better cognitive functioning
Change in cognitive functioning evaluated through MMSE | 13 weeks after the beginning of the intervention
  Cognitive functioning is assessed using the MMSE is a widely used screening tool that evaluates global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.

SECONDARY OUTCOMES:
Mood assessed through the Geriatric Depression Scale-15 (GDS-15) | baseline
  The GDS-15 is used to measure mood. It is considered a reliable tool to screen depressive symptoms in older people. With a dichotomous format (yes/no answers), this scale assesses depression in older people. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
Change in mood assessed through the GDS-15 | 13 weeks after the beginning of the intervention
  The GDS-15 is used to measure mood. It is considered a reliable tool to screen depressive symptoms in older people. With a dichotomous format (yes/no answers), this scale assesses depression in older people. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
Anxiety symptomatology assessed through the Geriatric Anxiety Inventory (GAI) | baseline
  It assesses, in several contexts, the severity of anxiety symptoms in the older adults. It consists in 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Change in anxiety symptomatology assessed through the GAI | 13 weeks after the beginning of the intervention
  It assesses, in several contexts, the severity of anxiety symptoms in the older adults. It consists in 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Quality of life evaluated through Quality of Life - Alzheimer's Disease (QoL-AD) | baseline
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.
Change in quality of life evaluated through QoL-AD | 13 weeks after the beginning of the intervention
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.
Quality of life evaluated through dementia Quality of Life scale (DEMQoL) | baseline
  The DEMQoL is used to assess quality of life. Suitable for use in cases of mild/moderate dementia (MMSE score higher or equal 10 points) based on information provided by the patient (patient version). This 29-item scale assesses perceptions of daily activities and looking after yourself, health and well-being, cognitive functioning, social relationships and self-concept. The first 28 items are summed to calculate the DEMQOL score. Scores range from 28 to 112,with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.
Change in quality of life evaluated through DEMQoL | 13 weeks after the beginning of the intervention
  The DEMQoL is used to assess quality of life. Suitable for use in cases of mild/moderate dementia (MMSE score higher or equal 10 points) based on information provided by the patient (patient version). This 29-item scale assesses perceptions of daily activities and looking after yourself, health and well-being, cognitive functioning, social relationships and self-concept. The first 28 items are summed to calculate the DEMQOL score. Scores range from 28 to 112,with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.

OTHER OUTCOMES:
Sociodemographic information gathered through the sociodemographic questionnaire | baseline
  Participants' answers in the sociodemographic questionnaire designed specifically for this study. It gathers information about age, gender, educational level, marital status, type of institution attended, and clinical condition and will be administered to all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I. Justo Henriques, PhD, Study Director — Polytechnic University of Beja; Célia C Silva, BsC, Principal Investigator — Polytechnic University of Beja
Locations (4):
- Portugal (4):
  - Centro Social e Paroquial de Brinches, Serpa, Beja District
  - Centro Social Remelhe D. António Barroso, Barcelos, Braga District
  - Associação de Socorros da Freguesia Turcifal, Torres Vedras, Lisbon District
  - Fundação João Bento Raimundo, Guarda

IPD SHARING:
Plan to Share IPD: No